CLINICAL TRIAL: NCT02165514
Title: Traditional Cobb Angle Measurement of Kyphosis and Scoliosis Using Lunar IDXA
Brief Title: Cobb Angle Measurement of Kyphosis and Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Yebin Jiang, M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00029355
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Kyphosis; Scoliosis
Keywords: spinal curvatures
MeSH Terms: conditions — Kyphosis; Scoliosis; Spinal Curvatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lunar iDXA (DEXA) scan (Experimental): Spinal scans taken by DEXA scanner
  Interventions: Procedure: Lunar iDXA x-ray scan

INTERVENTIONS:
Procedure: Lunar iDXA x-ray scan — Subjects will lay either on their back or side depending whether subject has kyphosis or scoliosis. After the DEXA scan the computer will calculate the Cobb angle. The calculation of Cobb angle from the DEXA scan will be compared to the conventional spine x-ray.

SUMMARY:
Measurement of bone length in subjects diagnosed with kyphosis and scoliosis using the Lunar iDXA x-ray scan.

DETAILED DESCRIPTION:
To determine if bone density scanning (DEXA) and the use of a computer software program can make accurate measurements of the curvature(s) of the spine (Cobb angle)in patients with kyphosis and scoliosis compared to x-rays of the spine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Have Kyphosis or Scoliosis
* Have had an x-ray of the spine performed within 3 months time

Exclusion Criteria:

* Are unwilling to read and sign this document
* Are pregnant or if you have not had a negative pregnancy test just prior to the iDXA scan.
* Have severe deformities of your back
* Unable to lay on the scanning table for the scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cobb angle measurements in degrees of spine curvature | 3 year
  Comparison of iDXA Cobb anle measurements with Cobb angle measurements from radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Yebin Jiang, PhD, Principal Investigator — University of Michigan Hospital